CLINICAL TRIAL: NCT01143987
Title: Effect of Cinacalcet Treatment on Vascular Arterial Stiffness Among Peritoneal Dialysis Patients With Secondary Hyperparathyroidism
Brief Title: Cincalcet and Vascular Arterial Stiffness Among Peritoneal Dialysis Patients With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chow Kai Ming, Associate Consultant, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2010.084-T
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Hyperparathyroidism; Arterial Stiffness
Keywords: hyperparathyroidism; pulse wave velocity; end-stage renal disease; arterial stiffness
MeSH Terms: conditions — Hyperparathyroidism; Kidney Failure, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cinacalcet (Experimental): Oral cinacalcet
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — starting with 25 mg daily dose with titration, maximum dose 100 mg daily
  Other Names: Sensipar

SUMMARY:
Active parathyroid glands among renal dialysis patients contribute to calcified and hardened blood vessels. Such damage to the blood vessels, in turn, takes a significant toll in terms of cardiovascular disease. Calcimimetics has been suggested to lower the risk of vascular calcification. Role of cinacalcet was demonstrated in animal model but human data are lacking. The investigators designed an open label pilot study to evaluate the effect of cinacalcet in 20 peritoneal dialysis patients with inadequately controlled secondary hyperparathyroidism despite standard treatment. The primary outcome is the aortic pulse wave velocity at 26 and 52 months after cinacalcet treatment.

DETAILED DESCRIPTION:
Mineral metabolism disturbance and hyperparathyroidism contribute to arterial stiffness and vascular calcification. The vascular damage, in turn, contributes to significant cardiovascular morbidity and mortality of end-stage renal disease patients. Calcimimetics has been suggested to lower the risk of vascular calcification. Role of cinacalcet was demonstrated in animal model but human data are lacking. We design an open label pilot study to evaluate the effect of cinacalcet in 20 peritoneal dialysis patients with inadequately controlled secondary hyperparathyroidism despite standard treatment. The primary outcome is the aortic pulse wave velocity at 26 and 52 months after cinacalcet treatment.

ELIGIBILITY:
Inclusion Criteria:

* plasma parathyroid hormone level of at least 300 pg/ml (31.8 pmol/L)
* aged 18 or older on peritoneal dialysis for at least three months
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* evidence of cancer, active infection or diseases with limited life expectancy
* diseases known to cause hypercalcaemia
* adjusted serum calcium level below 2.1 mmol/L (8.4 mg/dL) after correction for albumin
* participation in another interventional study within last 30 days of randomization
* history of a psychological illness or condition that would interfere with the patient's ability to understand the requirement of the study and/or comply with the study procedures
* patients receiving drugs with a narrow therapeutic index and metabolized by cytochrome P-450 2D6 (which is inhibited by cinacalcet): flecainide, thioridazine and most tricyclic antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Aortic pulse wave velocity after the cinacalcet treatment | change in aortic pulse wave velocity at 52 weeks from baseline
  as before

SECONDARY OUTCOMES:
Percent change in the values for parathyroid hormone levels | within one year of treatment with cinacalcet
  Blood samples will be stored before and after treatment with cinacalcet for further analysis.
Change in calcium levels | within one year of treatment with cinacalcet
  as before
Aortic pulse wave velocity after the cinacalcet treatment | change in aortic pulse wave velocity at 26 weeks from baseline
  as stated in the description of Primary Outcome Measure
Change in phosphorus levels | within one year of cinacalcet treatment
  as before
Change in calcium-phosphorus product | within one year of cinacalcet treatment
  as before

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ming Chow, MBChB, Principal Investigator — Chinese University of Hong Kong, Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

REFERENCES:
- [Derived] Chow KM, Szeto CC, Kwan BC, Cheng PM, Pang WF, Leung CB, Li PK. Effect of cinacalcet treatment on vascular arterial stiffness among peritoneal dialysis patients with secondary hyperparathyroidism. Nephrology (Carlton). 2014 Jun;19(6):339-44. doi: 10.1111/nep.12223. PMID 24589316